CLINICAL TRIAL: NCT00604461
Title: Phase I/II Trial of Carboplatin, Bevacizumab and Pemetrexed in the First-Line Treatment of Patients With Malignant Pleural Mesothelioma (MPM)
Brief Title: Carboplatin, Bevacizumab and Pemetrexed in the First-Line Treatment of Patients With Malignant Pleural Mesothelioma (MPM)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14896; AVF3483s (Other: Genentech)
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Results first posted 2011-12-26 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2011-11

CONDITIONS: Mesothelioma
Keywords: Carboplatin; Bevacizumab; Avastin; Pemetrexed; Alimta
MeSH Terms: conditions — Mesothelioma | interventions — Carboplatin; Bevacizumab; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose Escalation Followed by Maintenance Therapy (Experimental): A: Tiered Dose Escalation/Phase II Dose -
  * Tier -1: Carboplatin AUC 4 + Bevacizumab 15 mg/Kg+Pemetrexed 500 mg/m^2.
  * Tier 1: Carboplatin AUC 5 + Bevacizumab 15 mg/Kg+Pemetrexed 500 mg/m^2.
  * Tier 2: Carboplatin AUC 6 + Bevacizumab 15 mg/Kg+Pemetrexed 500 mg/m^2.
  B: Maintenance Therapy -
  * Patient was maintained on pemetrexed plus bevacizumab for a total of one year after initiation of maintenance or until progression which ever occured first.
  Interventions: Drug: Carboplatin, Bevacizumab and Pemetrexed

INTERVENTIONS:
Drug: Carboplatin, Bevacizumab and Pemetrexed — Chemotherapy was given for 2 cycles after maximal response. Patients were taken off study at the time of progression. If the patient had stable disease or better, as a response, then the patient was maintained on pemetrexed plus bevacizumab for a total of one year after initiation of maintenance or until progression which ever occured first. Computed tomography (CT) scans were be done every 12 weeks during the maintenance phase.
  Other Names: Bevacizumab (Avastin™); Pemetrexed (Alimta™)

SUMMARY:
The purpose of this research study was to evaluate how effective the combination of Carboplatin, Bevacizumab (Avastin™) and, Pemetrexed (Alimta™) is in the treatment of patients with Malignant Pleural Mesothelioma (MPM). A combination of cisplatin and pemetrexed is considered standard for this disease and typically off protocol patients would receive cisplatin or carboplatin and pemetrexed as standard of care.

The planned length of the study (first patient screened to last patient enrolled) was 24 months. The planned length of the entire study (enrollment period + the treatment period + a follow-up period of at least 12 months) was 36 months.

DETAILED DESCRIPTION:
This was a planned Phase I/II dose escalation study. Patients were enrolled in a cohort of 3.

Eligible patients with unresectable pleural mesothelioma received frontline treatment consisting of carboplatin AUC 5, bevacizumab 15 mg/kg, and pemetrexed 500 mg/m^2 every 21 days (Tier-1). Dose escalation continued to achieve a target dosage using carboplatin AUC 6 (Tier-2). After a maximum of 6 treatment cycles, non-progressing patients received maintenance therapy with bevacizumab and pemetrexed every 21 days to complete 1-year total treatment duration.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically proven diagnosis of Malignant Pleural Mesothelioma (MPM)
* Patient must have MPM with measurable disease.
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Patient must have adequate renal function with a serum creatinine level of less than 1.5 mg/dl and patient should have a calculated creatinine clearance of more than 40ml/min.
* Patient must have adequate hepatic function with a serum bilirubin level of less that 3mg/dl, and an alkaline phosphatase, ALT and AST of less than five times the upper limit of normal
* Patient must also have evidence of adequate bone marrow function with an absolute neutrophil count of more than 1500 cells per deciliter and a platelet count of more than 100,000 per deciliter.
* Patients must be more than 28 days since prior open biopsy; more than 7 days since prior fine-needle aspiration; more than 7 days since prior core biopsy; more than 28 days since prior surgery.
* Patients must be able to take dexamethasone, folic acid, and vitamin B-12 supplementation.
* All patients must sign informed consent that will detail the investigational nature of the study in accordance with the institutional and federal guidelines.
* Patients with clinically significant pleural effusions or ascites (symptomatic or detectable by clinical exam) should have their effusions drained prior to enrollment on the clinical trial.

Exclusion Criteria:

* Patients with hypercalcemia (corrected calcium of more than 11 mg/dl) will be excluded.
* Patients with history of hemoptysis, haematemesis, coagulopathy or thrombosis will be excluded.
* Patients requiring anticoagulation for any reason will be excluded.
* History of palliative radiation therapy within 2 weeks
* Blood pressure of >160/100 mmHg, despite adequate anti-hypertensive use.
* Currently ongoing unstable angina
* New York Heart Association (NYHA) Grade II or greater congestive heart failure.
* History of stroke within 6 months
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to the day of initiation of treatment, anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to the day of initiation of treatment.
* Pregnant (positive pregnancy test) or lactating
* Urine calculated creatinine clearance of less than 40ml/minute. - History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture
* Inability to comply with study and/or follow-up procedures

Laboratory Values:

* Patient must have adequate renal function with a serum creatinine level of less than 1.5 mg/dl and patient should have a calculated creatinine clearance of more than 40ml/min.
* Patient must have adequate hepatic function with a serum bilirubin level of less than 3 mg/dl, and an alkaline phosphatase, ALT and AST of less than five times the upper limit of normal
* Patient must also have evidence of adequate bone marrow function with an absolute neutrophil count of more than 1, 500 cells per deciliter and a platelet count of more than 100,000 per deciliter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tawee Tanvetyanon, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was Open to Accrual (recruiting) for a period of 2 years (10/04/07 through 10/05/09). Recruiting ended on 10/05/09 due to slow accrual, as requested by pharmaceutical company.
Groups:
- Dose Escalation Followed by Maintenance Therapy: A: Tiered Dose Escalation/Phase II Dose. Tier -1: Carboplatin AUC 4 + Bevacizumab 15 mg/Kg+Pemetrexed 500 mg/m^2. Tier 1: Carboplatin AUC 5 + Bevacizumab 15 mg/Kg+Pemetrexed 500 mg/m^2. Tier 2: Carboplatin AUC 6 + Bevacizumab 15 mg/Kg+Pemetrexed 500 mg/m^2.
  B: Maintenance Therapy - Patient was maintained on pemetrexed plus bevacizumab for a total of one year after initiation of maintenance or until progression which ever occured first.
Period: Overall Study
Arm/Group | Dose Escalation Followed by Maintenance Therapy
Started | 13
Completed | 12 (Death within 30 days of treatment occurred in 1 patient.)
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dose Escalation Followed by Maintenance Therapy
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 7
Age, Customized [Median (Full Range); unit: years] | 66 [41 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Partial Response (PR) of Target Lesions
Description: Tumor response was assessed in 12 patients who had at least one follow-up computed tomography (CT) scan. Response Evaluation Criteria in Solid Tumors (RECIST) definition of Partial Response: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 12 Months
Population: All participants with baseline and at least one post-baseline target lesion measurement.
Measure: Number; unit: participants
Arm/Group | Dose Escalation Followed by Maintenance Therapy
Number analyzed (Participants) | 12
participants | 4

2. Secondary Outcome: Number of Months of Progression Free Survival (PFS)
Description: The PFS is defined as the duration of time from the start of treatment to time of progression or death, whichever occurs first.
Time Frame: 2 Years, 9 Months
Population: All participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Escalation Followed by Maintenance Therapy
Number analyzed (Participants) | 13
Months | 7.8 [0 to 16.3]

ADVERSE EVENTS:
Time Frame: 2 Years, 9 MOnths
Arm/Group | Dose Escalation Followed by Maintenance Therapy
Serious Adverse Events (participants affected / at risk) | 4/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Followed by Maintenance Therapy (N=13)
Anemia (Blood and lymphatic system disorders) | 1 (1) — Grade 3
Death (General disorders) | 1 (1) — One patient died within 30 days of starting treatment from an unidentified cause.
Fatigue (General disorders) | 2 (2) — Grade 3
Infection (Infections and infestations) | 1 (1) — Grade 4
Leukopenia (Blood and lymphatic system disorders) | 1 (1) — Grade 3
Thromboembolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Followed by Maintenance Therapy (N=13)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anorexia (General disorders) | 4 (4)
Cardiac Arrhythmia (Cardiac disorders) | 1 (2)
Constipation/Diarrhea (Gastrointestinal disorders) | 5 (8)
Dysgeusia (General disorders) | 1 (1)
Elevated Creatinine (Renal and urinary disorders) | 1 (1)
Epistaxis (General disorders) | 2 (3)
Fatigue (Gastrointestinal disorders) | 9 (18)
Herpes Zoster (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 6 (8)
Mucositis (Gastrointestinal disorders) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 5 (11)
Pain (General disorders) | 8 (18)
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Transaminitis (Endocrine disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This trial was closed early due to slow patient accrual. The planned accrual had been 44.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No